CLINICAL TRIAL: NCT06127329
Title: Efficacy and Safety of Bronchial Infusion Chemotherapy Combined With Drug-loaded Microsphere Embolization of EqualSpheres in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of BAI Combined With DEB-BACE of EqualSpheres in the Treatment of Advanced NSCLC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gang Wu (Other)
Responsible Party: Sponsor-Investigator, Gang Wu, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-KY-1101-001
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAI combine with DEB-BACE (Experimental): Procedure: BAI combine with DEB-BACE: bronchial infusion chemotherapy combined with drug-loaded microsphere embolization of EqualSpheres
  1. First treatment. Only infusion chemotherapy (THP + Platinum + Letitrexed), THP 20 ~30mg/m2, Nedaplatin 40mg/m2, Letitrexed 3mg/m2.
  2. Second treatment. After infusionchemotherapy, EqualSpheres microsphere used for embolization: EqualSpheres microspheres (400 μm) 1tube was loaded and adsorbed THP (40 ~ 60mg/m2). End point of embolization: stagnation of blood flow in tumor feeding artery.
  Interventions: Procedure: BAI combine with DEB-BACE

INTERVENTIONS:
Procedure: BAI combine with DEB-BACE — 1. First treatment. Only infusion chemotherapy (THP + Platinum + Letitrexed), THP 20 ~30mg/m2, Nedaplatin 40mg/m2, Letitrexed 3mg/m2.
  2. Second treatment. After infusionchemotherapy, EqualSpheres microsphere used for embolization: EqualSpheres microspheres (400 μm) 1tube was loaded and adsorbed THP (40 ~ 60mg/m2). End point of embolization: stagnation of blood flow in tumor feeding artery.

SUMMARY:
This is a prospective, single-arm, open-label study designed to evaluate the efficacy and safety of bronchial infusion chemotherapy（BAI） combined with drug-loaded microsphere embolization of EqualSpheres in advanced Non-small cell lung cancer (NSCLC). Progression-free survival (PFS) will be evaluated as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old, male and female;
2. According to the Guidelines for the Diagnosis and Treatment of Primary Lung Cancer (2022 edition), the patient was diagnosed with NSCLC by imaging and histopathology;
3. TNM stages were III-IV;
4. Newly diagnosed, first-line treatment failure, refusal or inability to perform conventional treatment (surgery, chemoradiotherapy);
5. ECOG PS ≤2;
6. Expected survival > 3 months;
7. Sign the informed consent voluntarily, and the compliance is good.

Exclusion Criteria:

1. Previously received interventional therapy (iodine particle implantation, ablation, TACE treatment);
2. Combined with extensive and uncontrolled extrapulmonary metastases, such as liver metastasis, bone metastasis, and brain metastasis;
3. Have had or currently having other primary malignant tumors;
4. White blood cell < 3×109/L, platelet count < 50×109/L, HGB < 90 g/L;
5. Hepatic and renal insufficiency (creatinine > 2 mg/L; AST and/or ALT > 2 times the normal upper limit);
6. Coagulation dysfunction (INR > 1.5) or known bleeding disease (except lung cancer combined with hemoptysis), or anticoagulation therapy;
7. Patients with active infection requiring antibiotic treatment;
8. Uncontrolled hypertension, diabetes, and cardiovascular disease with obvious symptoms;
9. contrast agent allergy;
10. Women with pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
ORR | up to 3 years
  ORR is defined as the percentages of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria
Overall survival (OS) | up to 3 years
  The time from recruitment to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Gang Wu, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No